CLINICAL TRIAL: NCT02432209
Title: Improving Reproductive Fitness Through Pretreatment With Lifestyle Modification in Obese Women With Unexplained Infertility
Acronym: FIT-PLESE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Penn State University (Other); Augusta University (Other); University of California, San Francisco (Other); University of North Carolina (Other); University of Oklahoma (Other); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIT-Plese
Record Dates: First submitted 2015-03-16; First posted 2015-05-04 (Estimated); Results first posted 2021-03-15 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — Caloric Restriction; Orlistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive Lifestyle Mod. Intervention (Active Comparator): The intensive lifestyle modification intervention will consist of caloric restriction (consumption of approximately 1200-1500 kcal/d), use of an over-the-counter weight loss medication (Alli, which is brand name Orlistat, a gastric lipase inhibitor that limits gut fat absorption), and moderate physical activity (goal of reaching 10,000 steps a day). The pretreatment intervention will last 16 weeks and is designed to promote a weight loss of approximately 7% of total body weight.
  Interventions: Other: Caloric Restriction; Drug: Orlistat; Other: Moderate physical activity
- Standard Lifestyle Intervention (Placebo Comparator): Women in the standard lifestyle intervention (standard) will receive publicly available written materials that promote engagement in moderate physical activity with target of 10,000 steps a day. Detailed instruction of physical activity will not be provided.
  Interventions: Other: Moderate physical activity

INTERVENTIONS:
Other: Caloric Restriction — Subjects on Active comparator will have Caloric Restriction to a 1200-1500 kcal/day diet through use of Nutrisystem Meal Plan.
  Other Names: Nutrisystem
  Arms: Intensive Lifestyle Mod. Intervention
Drug: Orlistat — Subjects on Active comparator will use an over-the-counter weight loss medication, Orlistat, a gastric lipase inhibitor that limits gut fat absorption.
  Other Names: Alli
  Arms: Intensive Lifestyle Mod. Intervention
Other: Moderate physical activity — All subjects in both arms will be encouraged to engage in moderate physical activity with target of 10,000 steps a day.

SUMMARY:
A two-arm, multicenter, prospective, randomized clinical trial of a lifestyle modification program with tracked increased physical activity and weight loss (intensive) compared to recommendations to tracking of increased physical activity alone with weight maintenance (standard) in women with obesity and unexplained infertility. This 16 week period of lifestyle modification will be followed by an open label empiric infertility treatment regimen consisting of three cycles of ovarian stimulation with oral medication (clomiphene citrate (CC)), triggering of ovulation with human chorionic gonadotropin (hCG) and intrauterine insemination (IUI).

DETAILED DESCRIPTION:
Study Objective An intensive lifestyle modification intervention (which includes caloric restriction, use of an over-the-counter weight loss medication, and moderate physical activity with tracking) designed to promote a weight loss of approximately 7% of initial body weight is more likely to achieve a good perinatal outcome (i.e. a healthy term normal weight infant) than a recommendation to standard lifestyle modification with moderate physical activity with tracking (based on publically available activity recommendations) in obese women with unexplained infertility.

Patient Population The population will consist of 380 obese women with unexplained infertility, age 18-40 years old. Subjects must have normal ovulatory function and normal ovarian reserve. Additionally, the couple will have no other major infertility factor: the subject will have at least one patent fallopian tube and a normal uterine cavity, and a partner total motile sperm count of at least 5 million in at least one ejaculate.

Study Design This will be a two-arm, multicenter, prospective, randomized clinical trial of a lifestyle modification program with tracked increased physical activity and weight loss (intensive) compared to recommendations to tracking of increased physical activity alone with weight maintenance (standard) in women with obesity and unexplained infertility. This 16 week period of lifestyle modification will be followed by an open label empiric infertility treatment regimen consisting of three cycles of ovarian stimulation with oral medication (clomiphene citrate (CC)), triggering of ovulation with human chorionic gonadotropin (hCG) and intrauterine insemination (IUI).

Treatment The intensive lifestyle modification intervention will consist of caloric restriction (consumption of approximately 1200-1500 kcal/d), use of an over-the-counter weight loss medication (Alli, which is brand name Orlistat, a gastric lipase inhibitor that limits gut fat absorption), and moderate physical activity (goal of reaching 10,000 steps a day). The pretreatment intervention will last 16 weeks and is designed to promote a weight loss of approximately 7% of total body weight. Women in the standard lifestyle intervention (standard) will receive publicly available written materials that promote engagement in moderate physical activity with target of 10,000 steps a day. Detailed instruction of physical activity will not be provided. Participants in both groups will receive activity tracking devices (Fitbit Wireless Activity Tracker) and wireless scales (Fitbit Aria Wireless Activity Scale) to promote adherence to the inventions and to allow monitoring for compliance by study personnel. The pretreatment intervention will last 16 weeks. Both groups will aim for activity levels of 10,000 steps/day, with a recommendation to increase steps from baseline by 500 steps/per week. The investigators will monitor subjects monthly during this preconception intervention. After 16 weeks of lifestyle modification, all subjects randomized will receive a standardized empiric infertility treatment, regardless of adherence or success in achieving treatment goals. This treatment will consist of ovarian stimulation with CC followed by ultrasound follicular monitoring, hCG trigger of ovulation, and a single partner intrauterine insemination (IUI) per treatment cycle for up to three treatment cycles. The goal for both treatment groups will be to maintain levels of physical activity and weight achieved during the pretreatment phase during the empiric infertility treatment phase. Subjects who conceive will be followed throughout pregnancy with the wireless activity monitor and wireless scale. Additionally there will be three brief onsite visits during pregnancy (per trimester at 16, 24, and 32 weeks) for onsite determination of weight, glycemic, and blood pressure changes and collection of biospecimens. All pregnancy outcomes will be tracked. Subjects who deliver will be encouraged to donate placenta and cord blood to the study repository and then to enroll in our Pregnancy Registry for continued infant follow-up. The investigators will also expand the number and variety of specimens that are collected for the repository from both partners including urine and serum, semen, saliva, placenta and cord blood.

ELIGIBILITY:
Inclusion Criteria:

1. Women ≥18 to ≤ 40 years of age, with one or more years infertility history, desirous of conceiving, regularly ovulating (defined as 9 or more menses per year), at initiation of participation.
2. BMI ≥ 30 kg/m2.
3. Normal uterine cavity and at least one open fallopian tube confirmed by hysterosalpingography (HSG), sonohysterography (SHG), or laparoscopy/hysteroscopy in the last three years preceding enrollment into the study. An uncomplicated intrauterine non-IVF pregnancy and uncomplicated delivery and postpartum course resulting in live birth within the last three years will also serve as sufficient evidence of a patent tube and normal uterine cavity as long as the subject did not have, during the pregnancy or subsequently, risk factors for Asherman's syndrome or serious pelvic infection or other disorder leading to an increased suspicion for intrauterine abnormality or tubal occlusion.
4. Evidence of ovarian function/reserve as assessed by menstrual cycle day 3 (+/-2 days) FSH ≤10 IU/L with estradiol ≤ 70 pg/mL OR AMH ≥ 1 ng/mL within one year prior to study initiation.
5. Normal or corrected thyroid function within one year of study initiation.
6. Normal or corrected prolactin level within one year of study initiation.
7. In general good health, not taking any medications which could interfere with the study (e.g., FSH, insulin sensitizers).
8. Ability to have inseminations following hCG administration.
9. Male partner with total motile sperm in the ejaculate of at least 5 million sperm, within one year of study initiation.
10. Able to comply with intercourse instructions and collection of semen for insemination.

Exclusion Criteria:

1. Currently pregnant or successful pregnancies within 12 months of initiating participation. Clinical intrauterine miscarriages prior to initiating participation, within ASRM guidelines: subjects over 35 must wait six months, while subjects under 35 must wait 12 months. No exclusion for biochemical pregnancies.
2. Undiagnosed abnormal uterine bleeding.
3. Suspicious ovarian mass.
4. Subjects on oral contraceptives, depo-progestins, or hormonal implants (including Implanon). A two month washout period will be required prior to screening for patients on these agents. Longer washouts may be necessary for certain depot contraceptive methods or implants, especially when the implants are still in place. A one-month washout will be required for patients taking oral cyclic progestins.
5. Known 21-hydroxylase deficiency or other enzyme defect causing congenital adrenal hyperplasia.
6. Type I or Type II diabetes mellitus, or if receiving antidiabetic medications.
7. Known significant anemia (Hemoglobin <10 g/dL).
8. History of deep venous thrombosis, pulmonary embolus, or cerebrovascular event.
9. Known heart disease (New York Heart Association Class II or higher).
10. Known Liver disease (defined as AST or ALT>2 times normal, or total bilirubin >2.5 mg/dL).
11. Known Renal disease (defined as BUN >30 mg/dL or serum creatinine > 1.4 mg/dL).
12. History of, or suspected cervical carcinoma, endometrial carcinoma or breast carcinoma.
13. History of alcohol abuse (defined as >14 drinks/week) or binge drinking of ≥ 6 drinks at one time).
14. Known Cushing's disease.
15. Known or suspected adrenal or ovarian androgen secreting tumors.
16. Allergy or contraindication to the treatment medications: CC or hCG.
17. Couples with previous sterilization procedures (e.g. vasectomy, tubal ligation) whether or not it has been reversed.
18. Subjects with untreated poorly controlled hypertension defined as a systolic blood pressure ≥ 160 mm Hg or a diastolic ≥ 100 mm Hg obtained on two measures at least 60 minutes apart.
19. Subjects who have undergone a bariatric surgery procedure in the past or are in a period of acute weight loss (defined as a weight loss of greater than 5 kgs in the last 6 months).
20. Known moderate or severe endometriosis.
21. Anovulation or oligo-ovulation including hypothalamic amenorrhea, polycystic ovary syndrome, etc.
22. Donated semen.
23. Couples in which either partner is legally married to someone else.
24. Medical conditions that are contraindications to pregnancy.
25. Presence of severe, untreated psychiatric illness (major depression, substance abuse, eating disorder, etc.) that would, in the opinion of the site investigator, interfere with the patient's ability to successfully complete the study.
26. Any additional medical conditions that would be a contraindication to orlistat. (This includes patients with chronic malabsorption syndrome or cholestasis or known hypersensitivity to any of the drugs used in this study.)
27. Any contraindication to study requirements including diet recommendations and activity requirements.
28. Currently participating in a lifestyle intervention program (such as Weight Watchers, Atkins Diet, Curves) or lost more than 5% body weight within the last 6 months.
29. History of Gout.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 379 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nanette Santoro, MD, Study Chair — University of Colorado, Denver; Heping Zhang, PhD, Study Director — Yale University; Richard Legro, MD, Principal Investigator — Penn State University; Michael Diamond, MD, Study Director — Augusta University; Marcelle Cedars, MD, Study Director — University of California, San Francisco; Anne Steiner, MD MPH, Study Director — Univeristy of North Carolina; Karl Hansen, MD PhD, Study Director — University of Oklahoma; Christos Coutifaris, MD PhD, Study Director — University of Pennsylvania; Esther Eisenberg, MD MPH, Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (10):
- United States (10):
  - University of California San Francisco, San Francisco, California
  - Augusta University, Augusta, Georgia
  - Wayne State University, Southfield, Michigan
  - University of Rochester, Rochester, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Atrium Health Carolinas Healthcare System, Charlotte, North Carolina
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Pennsylvania State University, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with other researchers through the NICHD DASH system. It will be available 6 months after publication of the primary results.

REFERENCES:
- [Derived] Vitek WS, Sun F, Cardozo E, Hoeger KM, Hansen KR, Santoro N, Zhang H, Legro RS. Moderate and increased physical activity is not detrimental to live birth rates among women with unexplained infertility and obesity. F S Rep. 2023 Jun 24;4(3):308-312. doi: 10.1016/j.xfre.2023.06.004. eCollection 2023 Sep. PMID 37719091
- [Derived] Legro RS, Hansen KR, Diamond MP, Steiner AZ, Coutifaris C, Cedars MI, Hoeger KM, Usadi R, Johnstone EB, Haisenleder DJ, Wild RA, Barnhart KT, Mersereau J, Trussell JC, Krawetz SA, Kris-Etherton PM, Sarwer DB, Santoro N, Eisenberg E, Huang H, Zhang H; Reproductive Medicine Network. Effects of preconception lifestyle intervention in infertile women with obesity: The FIT-PLESE randomized controlled trial. PLoS Med. 2022 Jan 18;19(1):e1003883. doi: 10.1371/journal.pmed.1003883. eCollection 2022 Jan. PMID 35041662

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intensive Lifestyle Mod. Intervention | Standard Lifestyle Intervention
Started | 188 | 191
Completed | 157 | 151
Not Completed | 31 | 40

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensive Lifestyle Mod. Intervention | Standard Lifestyle Intervention | Total
Number analyzed (Participants) | 188 | 191 | 379
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 32 [29 to 35] | 32 [30 to 35] | 32 [29 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 188 | 191 | 379
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 9 | 12
  Not Hispanic or Latino | 179 | 177 | 356
  Unknown or Not Reported | 6 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 45 | 37 | 82
  White | 126 | 140 | 266
  More than one race | 6 | 5 | 11
  Unknown or Not Reported | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Rate of Good Birth Outcomes
Description: Defined as a live birth of an infant born at ≥ 37 weeks, with a birth weight between 2500 and 4000g and without a major congenital anomaly
Time Frame: At time of birth, approximately 17 months into the study
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Lifestyle Mod. Intervention | Standard Lifestyle Intervention
Number analyzed (Participants) | 188 | 191
Participants | 23 | 29
Statistical Analysis 1: Comparison: Intensive Lifestyle Mod. Intervention vs Standard Lifestyle Intervention; Test type: Superiority; p = 0.404, Chi-squared; Risk Ratio (RR) = 0.81, 95% CI 2-sided [0.48 to 1.34]

2. Secondary Outcome: Live Birth Rate
Description: All the live birth for the study
Time Frame: At time of birth, approximately 17 months into the study
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Lifestyle Mod. Intervention | Standard Lifestyle Intervention
Number analyzed (Participants) | 188 | 191
Participants | 38 | 42

3. Secondary Outcome: Time to Pregnancy in Days
Description: Days from randomization to the first known date of conception
Time Frame: 0-8 months
Population: For those who achieved pregnancy
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Intensive Lifestyle Mod. Intervention | Standard Lifestyle Intervention
Number analyzed (Participants) | 59 | 52
days | 160 [102 to 190] | 163 [98.5 to 214]

4. Secondary Outcome: Pregnancy Loss Rate
Description: Pregnancy loss (conception without a live birth) among those who achieved pregnancy
Time Frame: After conception, 0-13 months into the study
Population: For those who achieved pregnancy
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Lifestyle Mod. Intervention | Standard Lifestyle Intervention
Number analyzed (Participants) | 63 | 59
Participants | 24 | 14

5. Secondary Outcome: Multiple Pregnancy Rate
Description: Determined by number of multiple pregnancies / number of pregnancies
Time Frame: After conception, 1-13 months into the study
Population: For those with clinical pregnancy
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Lifestyle Mod. Intervention | Standard Lifestyle Intervention
Number analyzed (Participants) | 48 | 45
Participants | 7 | 3

6. Secondary Outcome: Birth Weight in Grams
Description: Birth weight (grams) for infant delivered
Time Frame: at time of birth, approximately 17 months into the study
Population: For the live-born infants
Measure: Median (Inter-Quartile Range); unit: gram
Arm/Group | Intensive Lifestyle Mod. Intervention | Standard Lifestyle Intervention
Number analyzed (Participants) | 36 | 42
gram | 3217.7 [2802.4 to 3642.9] | 3189.3 [2636.5 to 3671.3]

7. Secondary Outcome: Mode of Delivery-Cesarean Section
Description: Babies by Cesarean Section/Number of participants who delivered baby
Time Frame: At time of birth, approximately 17 months into the study
Population: For those who delivered baby(babies)
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Lifestyle Mod. Intervention | Standard Lifestyle Intervention
Number analyzed (Participants) | 36 | 40
Participants | 19 | 23

ADVERSE EVENTS:
Time Frame: From randomization to 6 weeks following infant delivery (from 0 to up to 18.5 months)
Arm/Group | Intensive Lifestyle Mod. Intervention | Standard Lifestyle Intervention
All-Cause Mortality (participants affected / at risk) | 0/188 | 0/191
Serious Adverse Events (participants affected / at risk) | 12/188 | 13/191
Other Adverse Events (participants affected / at risk) | 157/188 | 157/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Intensive Lifestyle Mod. Intervention (N=188) | Standard Lifestyle Intervention (N=191)
Hospitalization (Endocrine disorders) | 2 | 0
Pelvic pain (Endocrine disorders) | 1 | 0
Appendicitis (General disorders) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Complex cyst resulting in surgical intervention (General disorders) | 0 | 1
Hospitalization during first trimester (Pregnancy, puerperium and perinatal conditions) | 1/63 | 0/59 — For those who achieved pregnancy
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1/63 | 2/59 — For those who achieved pregnancy
Pregnancy of Unknown Location (Pregnancy, puerperium and perinatal conditions) | 3/63 | 3/59 — For those who achieved pregnancy
Marginal Placenta Previa (Pregnancy, puerperium and perinatal conditions) | 1/63 | 0/59 — For those who achieved pregnancy
Placenta Previa and Pre-term birth (Pregnancy, puerperium and perinatal conditions) | 0/63 | 1/59 — For those who achieved pregnancy
Hospitalization (General disorders) | 2/63 | 1/59 — For those who achieved pregnancy
Hospitalization-infant (Pregnancy, puerperium and perinatal conditions) | 1/38 | 2/42 — For the live-born infants
Myelomeningocele (Pregnancy, puerperium and perinatal conditions) | 1/38 | 0/42 — For the live-born infants
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Intensive Lifestyle Mod. Intervention (N=188) | Standard Lifestyle Intervention (N=191)
Constipation (Cardiac disorders) | 23 | 7
Diarrhea (General disorders) | 35 | 9
Fever (General disorders) | 5 | 0
Flatulence (Gastrointestinal disorders) | 33 | 2
Mood swings (General disorders) | 2 | 9
Nausea/vomiting (General disorders) | 41 | 24
Oily stools/discharge (Gastrointestinal disorders) | 43 | 0
Pre-term labor (Pregnancy, puerperium and perinatal conditions) | 2/63 | 6/59 — For those who achieved pregnancy
Pre-eclampsia/Eclampsia (Pregnancy, puerperium and perinatal conditions) | 4/63 | 7/59 — For those who achieved pregnancy
Gestational Diabetes (Pregnancy, puerperium and perinatal conditions) | 6/63 | 10/59 — For those who achieved pregnancy
Incompetent cervix (Pregnancy, puerperium and perinatal conditions) | 2/63 | 0/59 — For those who achieved pregnancy
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 2/63 | 4/59 — For those who achieved pregnancy
Placental abnormalities (Pregnancy, puerperium and perinatal conditions) | 5/63 | 4/59 — For those who achieved pregnancy
Post-partum Infection (Pregnancy, puerperium and perinatal conditions) | 0/63 | 2/59 — For those who achieved pregnancy
Post-partum hemorrhage (Pregnancy, puerperium and perinatal conditions) | 0/63 | 1/59 — For those who achieved pregnancy
Other complication (Pregnancy, puerperium and perinatal conditions) | 4/63 | 3/59 — For those who achieved pregnancy
Other post-partum complication(s) (Pregnancy, puerperium and perinatal conditions) | 3/63 | 1/59 — For those who achieved pregnancy
Intrauterine growth restriction (Pregnancy, puerperium and perinatal conditions) | 1/38 | 4/42 — For the live-born infants
Admission to NICU (Pregnancy, puerperium and perinatal conditions) | 7/38 | 12/42 — For the live-born infants
Abdominal pain (General disorders) | 20 | 12
Anxiety/irritability (General disorders) | 11 | 14
Back pain (General disorders) | 13 | 20
Dysmenorrhea (Reproductive system and breast disorders) | 23 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-07-03): https://cdn.clinicaltrials.gov/large-docs/09/NCT02432209/Prot_SAP_ICF_000.pdf